CLINICAL TRIAL: NCT03532438
Title: Whole Genome Sequencing of Nontuberculous Mycobacterium (NTM) Derived From Sputum Specimen of NTM Lung Disease Patients Living Together and From Their Environmental Samples
Brief Title: WGS of NTM From Sputum of NTM Lung Disease Patients and From Their Environments
Acronym: NTM_HOME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Joon Yim, Professor, Seoul National University Hospital
Other Study IDs: NTM_HOME
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Nontuberculous Mycobacterium Infection; Whole Genome Sequencing
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA extracts from NTM derived from the patients and their environments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NTM patient group: NTM lung disease patients living together

SUMMARY:
The purpose of the study is to identify the genetic closeness of NTM derived from patients living together and from their surrounding environment and to trace the temporal relationship between them.

DETAILED DESCRIPTION:
After NTM isolation is done by using culture, from patients' sputum/bronchoscopic samples and their environmental samples, whole genome sequencing (WGS) will be conducted for all NTM isolates. Phylogenetic analysis will be performed based on single nucleotide polymorphism (SNP) on each NTM.

ELIGIBILITY:
Inclusion Criteria:

* The adult over 18 years of age
* The patient who have respiratory symptoms consistent with NTM, such as a chronic cough, sputum, and hemoptysis, who have NTM-positive findings on CT, and who have NTM identification in two or more sputum cultures or in one or more bronchoscopic/tissue culture. (2007 ATS/IDSA guideline)
* Pairs of patients living in the same household since diagnosis on NTM lung disease
* Consent to a collection of environmental samples from the patient's residence.

Exclusion Criteria:

* If the patient does not agree or withdraw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the patients visiting Seoul National University Hospital outpatient clinic, pairs of adult NTM lung disease patients who living together at the time of diagnosis were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Genetic similarity of NTM(Non-Tuberculous Mycobacterium) | Baseline
  Concordance of Single Nucleotide Polymorphisms (SNP) from NTMs derived from patients and their environments

CONTACTS AND LOCATIONS:
Overall Officials: Jae-June Yim, MD, Principal Investigator — Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine
Locations (1):
- Division of Pulmonology and Critical Care Medicine, Department of Internal Medicine and Lung Institute of Medical Research Center, Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bryant JM, Grogono DM, Greaves D, Foweraker J, Roddick I, Inns T, Reacher M, Haworth CS, Curran MD, Harris SR, Peacock SJ, Parkhill J, Floto RA. Whole-genome sequencing to identify transmission of Mycobacterium abscessus between patients with cystic fibrosis: a retrospective cohort study. Lancet. 2013 May 4;381(9877):1551-60. doi: 10.1016/S0140-6736(13)60632-7. Epub 2013 Mar 29. PMID 23541540
- [Background] Fournier PE, Dubourg G, Raoult D. Clinical detection and characterization of bacterial pathogens in the genomics era. Genome Med. 2014 Nov 29;6(11):114. doi: 10.1186/s13073-014-0114-2. eCollection 2014. PMID 25593594
- [Background] Roach DJ, Burton JN, Lee C, Stackhouse B, Butler-Wu SM, Cookson BT, Shendure J, Salipante SJ. A Year of Infection in the Intensive Care Unit: Prospective Whole Genome Sequencing of Bacterial Clinical Isolates Reveals Cryptic Transmissions and Novel Microbiota. PLoS Genet. 2015 Jul 31;11(7):e1005413. doi: 10.1371/journal.pgen.1005413. eCollection 2015 Jul. PMID 26230489
- [Background] Bryant JM, Grogono DM, Rodriguez-Rincon D, Everall I, Brown KP, Moreno P, Verma D, Hill E, Drijkoningen J, Gilligan P, Esther CR, Noone PG, Giddings O, Bell SC, Thomson R, Wainwright CE, Coulter C, Pandey S, Wood ME, Stockwell RE, Ramsay KA, Sherrard LJ, Kidd TJ, Jabbour N, Johnson GR, Knibbs LD, Morawska L, Sly PD, Jones A, Bilton D, Laurenson I, Ruddy M, Bourke S, Bowler IC, Chapman SJ, Clayton A, Cullen M, Daniels T, Dempsey O, Denton M, Desai M, Drew RJ, Edenborough F, Evans J, Folb J, Humphrey H, Isalska B, Jensen-Fangel S, Jonsson B, Jones AM, Katzenstein TL, Lillebaek T, MacGregor G, Mayell S, Millar M, Modha D, Nash EF, O'Brien C, O'Brien D, Ohri C, Pao CS, Peckham D, Perrin F, Perry A, Pressler T, Prtak L, Qvist T, Robb A, Rodgers H, Schaffer K, Shafi N, van Ingen J, Walshaw M, Watson D, West N, Whitehouse J, Haworth CS, Harris SR, Ordway D, Parkhill J, Floto RA. Emergence and spread of a human-transmissible multidrug-resistant nontuberculous mycobacterium. Science. 2016 Nov 11;354(6313):751-757. doi: 10.1126/science.aaf8156. PMID 27846606